CLINICAL TRIAL: NCT00679302
Title: A Double Blinded Randomized Controlled Trial for the Management of Pediatric Community Acquired Skin Abscesses - To Treat or Not to Treat With Antibiotics
Brief Title: Utility of Trimethoprim-sulfamethoxazole Use in Skin Abscess Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14415
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2014-03

CONDITIONS: Skin Diseases, Infectious
Keywords: skin abscess; CA-MRSA
MeSH Terms: conditions — Skin Diseases, Infectious | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; aluminum hydroxide, magnesium hydroxide, drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo group (Placebo Comparator): Maalox and bitter mixture
  Interventions: Drug: Placebo group
- antibiotic group (Active Comparator): Trimethoprim-sulfamethoxazole suspension
  Interventions: Drug: Trimethoprim-sulfamethoxazole

INTERVENTIONS:
Drug: Trimethoprim-sulfamethoxazole — Participants were randomized to receive placebo or trimethoprim/sulfamethoxazole using a computer randomization program on the initial presentation. The placebo is a Maalox and tonic water combination that resembled the antibiotic in color, texture and taste. The antibiotic dose is a standard trimethoprim/sulfamethoxazole for bacterial infection (10-12mg trimethoprim/kg/day, with a maximum adult dose of 160mg trimethoprim/day, divided into two doses). The concentration of the liquid is 200mg sulfamethoxazole/40mg trimethoprim per 5mL. With a maximum dose of 160mg trimethoprim, this equates to 20mL.
  Other Names: Septra
  Arms: antibiotic group
Drug: Placebo group — Placebo (Maalox with simethicone and bitter mixture) suspension was dispensed to study participants who were block randomized to receive the placebo.
  Other Names: Maalox (with simethicone and bitter mixture)
  Arms: placebo group

SUMMARY:
The purpose of this study is to determine if antibiotics are required in the management of skin abscess following incision and drainage.

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled trial at an urban pediatric emergency department. Sample size (162) was based on a threshold equivalence of 7% (α = 0.05, power = 80%). Inclusion criteria were: non-toxic, immunocompetent, 3 months to 18 years old, English-speaking patients with clinical or ultrasound identified skin abscesses who were not on antibiotics. Patients were block randomized to receive placebo or trimethoprim/sulfamethoxazole following incision and drainage. Follow-up was a call at 2-3 days & a repeat visit or call at 10-14 days. Treatment failure was defined as: persistent erythema, tenderness, and/or draining lesions. New lesion was defined as: primary resolution with development of new lesion (furuncle, carbuncle or abscess) at a different location. Compliance was evaluated by the return of the study medication or by patient report.

ELIGIBILITY:
Inclusion Criteria:

* non-toxic patients
* immunocompetent patients
* 3 months to 18 years old
* English-speaking patients
* skin abscesses
* not on antibiotics

Exclusion Criteria:

* toxic patients
* immunocompromising co-morbidities
* less than 3 months old or older than 18 years of age
* non-english speaking
* on antibiotics

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2006-07; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Peter, MD, Study Director — St. Louis University
Locations (1):
- Cardinal Glennon Children's Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Pallin DJ, Egan DJ, Pelletier AJ, Espinola JA, Hooper DC, Camargo CA Jr. Increased US emergency department visits for skin and soft tissue infections, and changes in antibiotic choices, during the emergence of community-associated methicillin-resistant Staphylococcus aureus. Ann Emerg Med. 2008 Mar;51(3):291-8. doi: 10.1016/j.annemergmed.2007.12.004. Epub 2008 Jan 28. PMID 18222564
- [Background] Korownyk C, Allan GM. Evidence-based approach to abscess management. Can Fam Physician. 2007 Oct;53(10):1680-4. PMID 17934031
- [Background] Cohen PR. Community-acquired methicillin-resistant Staphylococcus aureus skin infections: implications for patients and practitioners. Am J Clin Dermatol. 2007;8(5):259-70. doi: 10.2165/00128071-200708050-00001. PMID 17902728
- [Background] Lee MC, Rios AM, Aten MF, Mejias A, Cavuoti D, McCracken GH Jr, Hardy RD. Management and outcome of children with skin and soft tissue abscesses caused by community-acquired methicillin-resistant Staphylococcus aureus. Pediatr Infect Dis J. 2004 Feb;23(2):123-7. doi: 10.1097/01.inf.0000109288.06912.21. PMID 14872177
- [Derived] Duong M, Markwell S, Peter J, Barenkamp S. Randomized, controlled trial of antibiotics in the management of community-acquired skin abscesses in the pediatric patient. Ann Emerg Med. 2010 May;55(5):401-7. doi: 10.1016/j.annemergmed.2009.03.014. Epub 2009 May 5. PMID 19409657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients >3months and <18 years old with skin abscesses who are not immunocompromised, or in 3rd trimester of pregnancy were approached to participate in the study, or allergic to trimethoprim/sulfamethoxazole.
Pre-assignment Details: Enrolled participants were only excluded from the trial before assignment to groups if they left the emergency department prior to receiving the medication/placebo and further instructions.
Period: Overall Study
Arm/Group | Placebo Group | Antibiotic Group
Started | 84 | 77
Completed | 76 | 73
Not Completed | 8 | 4
Not completed — Lost to Follow-up | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Antibiotic Group | Total
Number analyzed (Participants) | 84 | 77 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84 | 77 | 161
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.5 (0.5) | 4.5 (0.5) | 4.5 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 30 | 68
  Male | 46 | 47 | 93
Region of Enrollment [Number; unit: participants]
  United States | 84 | 77 | 161

OUTCOME MEASURES:

1. Primary Outcome: Skin Abscess Resolution
Time Frame: 10-14 days
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Placebo Group | Antibiotic Group
Number analyzed (Participants) | 76 | 73
participants | 4 [1.2 to 6.8] | 3 [1.2 to 6.8]

2. Secondary Outcome: New Lesion Development and Spread of Skin Abscesses (on Subject)
Description: The secondary outcomes of interest included the development of new lesions at a different site (>5cm away from original skin abscess) on day 10 clinical follow-up or self-report and 3 month telephone follow-up.
Time Frame: 10-14 days and 3 month
Measure: Number; unit: participants
Arm/Group | Placebo Group | Antibiotic Group
Number analyzed (Participants) | 52 | 46
participants | 15 | 13

ADVERSE EVENTS:
Description: Participants were called 2-3 days later to set up follow up at day 10-14 and enquiries are made regarding any medication side effects. Phone calls were made 3 months later for further follow ups on recurrences and if other family members had developed skin abscesses.
Arm/Group | Placebo Group | Antibiotic Group
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/73
Other Adverse Events (participants affected / at risk) | 7/76 | 13/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=76) | Antibiotic Group (N=73)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) — any rash other than a pustule, folliculitis, carbuncle or skin abscess
diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
vomiting and diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
bad taste (General disorders) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
Small sample size with large number of loss to follow up at the 3 month mark.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes